CLINICAL TRIAL: NCT00619710
Title: A Multicenter, Randomized, Double Blind, Comparative Trial of Intravenous MERREM (Meropenem, ICI 194,660) vs PRIMAXIN I.V. (Imipenem-cilastatin) in the Treatment of Hospitalised Subjects With Complicated Skin and Skin Structure Infections.
Brief Title: Complicated Skin and Skin Structure Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3591IL/0079; D9211C00079
Record Dates: First submitted 2008-02-06; First posted 2008-02-21 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Skin Infection; Abscess; Cellulitis
Keywords: skin infections; MERREM; PRIMAXIN IV; complex abscess; perirectal abscess; wound infections; infected ischemic/diabetic ulcers; cellulitis; Meropenem; Imipenem-cilastatin
MeSH Terms: conditions — Cellulitis; Abscess; Wound Infection | interventions — Meropenem; Cilastatin, Imipenem Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Experimental): Meropenem
  Interventions: Drug: Meropenem
- 2 (Active Comparator): Imipenem-cilastatin
  Interventions: Drug: Imipenem-cilastatin

INTERVENTIONS:
Drug: Meropenem — Intravenous
  Other Names: Merrem
  Arms: 1
Drug: Imipenem-cilastatin — Intravenous
  Other Names: Primaxin
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate the non-inferiority of meropenem (Merrem) and imipenem in hospitalised subjects with complicated skin and skin structure infections.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are hospitalized males and females, aged 13 years or older, with clinical evidence of complicated skin and skin structure bacterial infection with material suitable for culture from 1 primary site of infections
* Within 72 hours before enrollment or at the time of enrollment, all subjects must provide an appropriate specimen for culture and susceptibility testing
* Subjects who have been given prior antibacterial therapy within 14 days of trial entry may be entered only if a culture is obtained showing persistence of a pathogen in blood or at the site of infection

Exclusion Criteria:

* Subjects with a known or suspected hypersensitivity to cephalosporins, penicillins, or carbapenems
* Subjects with a history of seizure disorders or subjects currently receiving antiepileptic medication
* Subjects with underlying infections or conditions which would interfere with evaluation of this study

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2001-02; Primary Completion 2003-12 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
The primary measure is clinical response after all antibacterial treatment is stopped). | 7-28 days

SECONDARY OUTCOMES:
clinical and microbiological response | Twice 3-28 days